CLINICAL TRIAL: NCT03860155
Title: An Interventional, Single Arm, Multicenter, Phase I/IIa Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-ACLF for the Treatment of Acute-on-Chronic Liver Failure (ACLF)
Brief Title: Allogeneic ABCB5-positive Stem Cells for Treatment of Acute-on-Chronic Liver Failure
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Very slow recruitment of patients and the current COVID-19 pandemic situation.
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Ticeba GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: allo-APZ2-ACLF-II-01
Record Dates: First submitted 2019-01-31; First posted 2019-03-01 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-09

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: Acute-on-Chronic Liver Failure; ACLF; ABCB5; ATP Binding Cassette Subfamily B Member 5; allogeneic; mesenchymal stem cells; advanced therapy medicinal product; somatic cell therapy; phase I/IIa
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- allo-APZ2-ACLF (Experimental): Application of IMP into peripheral vein (arm) by use of a perfusor.
  Interventions: Biological: allo-APZ2-ACLF

INTERVENTIONS:
Biological: allo-APZ2-ACLF — Administration of 2 x 10e6 allogeneic ABCB5-positive stem cells/kg bodyweight, each at Day 0, Day 5 (±1) and Day 13 (±1) into peripheral vein (arm) intravenously with a flow rate of 1-2 ml/min. Infusion of the product via a central venous catheter (CVC), a Port-a-Cath (Port) or a similar catheter is also possible. Allo-APZ2-ACLF will be in a concentration of 1 x 10e7 cells/mL in Human Serum Albumin/Ringer-Lactate/Glucose (HRG)-solution.
  Other Names: Skin-derived ABCB5-positive mesenchymal stem cells

SUMMARY:
This is an interventional, single arm, multicenter, phase I/IIa clinical trial. The study objective is to investigate the efficacy and safety of three i.v. doses of the investigational medicinal product (IMP) allo-APZ2-ACLF for the treatment of acute-on-chronic liver failure (ACLF). The allogeneic IMP allo-APZ2-ACLF contains skin-derived ABCB5-positive mesenchymal stem cells isolated from skin tissue of healthy donors and stored in a donor cell bank.

DETAILED DESCRIPTION:
This is an interventional, phase I/IIa clinical trial to investigate the efficacy (by changes in Model for End-Stage Liver Disease [MELD] score) and safety (by monitoring adverse events) of the IMP in patients with acute-on-chronic liver failure grade 2 and 3. The allogeneic IMP allo-APZ2-ACLF contains skin-derived ABCB5-positive mesenchymal stem cells isolated from skin tissue of healthy donors and stored in a donor cell bank.

The clinical trial will be conducted in Germany and will consist of a screening, treatment and efficacy follow-up period, and a safety follow-up period.The total duration is planned to be about 3 years including the follow-up period.

The planned sample size is up to 18 treated patients. 2 x 10e6 cells/kg, each at Day 0, Day 5 (±1) and Day 13 (±1), will be administrated into peripheral vein (arm) by use of a perfusor. allo-APZ2-ACLF will be in a concentration of 1 x 10e7 cells/mL in HRG-solution. In patients which require dialysis, the IMP application has to be performed at least 3 hours after end of dialysis. This is necessary to ensure that cells and secreted molecules are not cleared from the system by the dialysis.

Patients will be followed up for 24 weeks with clinic visits at Weeks 3, 4, 8, 12, 16, 20 and 24 after IMP application. Further safety follow-ups will be scheduled as home interviews via telephone at Months 15 and 24. If necessary (at the discretion of the investigator), safety follow-ups at Months 15 and 24 can also be carried out as an on-site visit.

The first six patients will be enrolled into the clinical trial consecutively with an interval of 2 weeks between the third IMP-application of the first patient and the enrolment of the second patient, etc. During this period the patient receives all three applications and immediate severe adverse effects (allergic reactions, SIRS) that could occur after treatment would be reported before treatment start of the next patient.

The safety data of these first six patients will be reviewed by the Medical Monitor continuously, if required with assistance of the further members of the DSMB. The safety evaluation of the DSMB will be submitted to the PEI and recruitment can only be continued after approval of an amendment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, aged 20 to 75 years;
2. Diagnosed ACLF of grade 2 or 3 according to EASL-CLIF definition;
3. Patients are not eligible for liver transplant (confirmed by transplantation board);
4. Histology result of liver biopsy not older than 4 weeks before screening;
5. Women of childbearing potential must have a negative blood pregnancy test at screening;
6. Women of childbearing potential and fertile men, and their partners must be willing to use highly effective contraceptive methods during the course of the clinical trial;
7. Written informed consent from patient, legal or authorized representative or a confirmation of justification of trial participation by an independent medical consultant. In case of confirmation by the independent medical consultant, a deferred informed consent from patient, legal or authorized representative has to be given.

Exclusion Criteria:

1. Patients without cirrhosis;
2. Patients with ACLF grade 1 according to EASL-CLIF definition;
3. Patient with septic shock;
4. Patients with known hepatopulmonal syndrome (HPS);
5. Patients with known pulmonary embolism that needs anticoagulative treatment;
6. Patients with pre-existing lung disease with necessity of respiratory support;
7. Active malignancy or history of malignancy within 5 years prior to trial entry;
8. Known infection with human immunodeficiency virus (HIV˗1, HIV-2);
9. Any known allergies to components of the IMP;
10. Current or previous (within 30 days of enrolment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
11. Patients anticipated to be unwilling or unable to comply with the requirements of the protocol;
12. Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
13. Pregnant or nursing women;
14. Employees of the sponsor, or employees or relatives of the investigator.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Change of Model for End-Stage Liver Disease (MELD) score at Week 24 or last available post-baseline measurement if the Week 24 score is missing. | Week 24, or last available post-baseline measurement of Days 5 (±1) or 13 (±1) or Weeks 3, 4, 8, 12, 16 or 20 if the Week 24 measurement is missing [LOCF].
  Model for End-Stage Liver Disease (MELD) score for assessing the severity of chronic liver disease is measured as absolute change to baseline score at Week 24 or last available post-baseline measurement if the Week 24 score is missing.
Assessment of adverse event (AE) occurrence | Between Screening and Month 24
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Change of MELD score at Weeks 3, 4, 8, 12, 16 and 20 | Weeks 3, 4, 8, 12, 16 and 20
  Model for End-Stage Liver Disease score is measured as absolute change to baseline score.
Change of Child-Pugh-Score at Weeks 3, 4, 8, 12, 16, 20 and 24 | Weeks 3, 4, 8, 12, 16, 20 and 24
  Child-Pugh-Score to assess the prognosis of chronic liver disease and cirrhosis is measured as absolute change to baseline score.
Change of CLIF-C ACLF score at Weeks 3, 4, 8, 12, 16, 20 and 24 | Weeks 3, 4, 8, 12, 16, 20 and 24
  CLIF-C ACLF score to assess the mortality in Acute-on-chronic liver failure patients is measured as absolute change to baseline score.
Overall survival time until Week 24 | Between Screening and Week 24
  Assessment of overall survival time.
Complications of ACLF (hepatorenal syndrome [HRS], variceal bleeding, ascites, hepatic encephalopathy [HE], spontaneous bacterial peritonitis [SBP]) | Between Screening and Week 24
  Assessment, documentation and evaluattion of ACLF related complications (hepatorenal syndrome, variceal bleeding, ascites, hepatic encephalopathy, spontaneous bacterial peritonitis).
Transient elastography assessment at Weeks 4, 12 and 24 | Weeks 4, 12 and 24
  Mapping of the elastic properties and the stiffness of the tissue as assessed by transient elastography imaging
Infections (proven infection necessitating systemic use of antibiotics) | Between Screening and Month 24
  All infections occurring during the clinical trial will be registered, documented and evaluated.
Change of levels of C-reactive protein in serum at Weeks 3, 4, 8, 12, 16, 20 and 24 | Weeks 3, 4, 8, 12, 16, 20 and 24
  C-reactive protein levels in the serum will be measured.
Liver Function Test (ALT, AST, AP, Albumin, Bilirubin, GGT) at Weeks 3, 4, 8, 12, 16, 20 and 24 | Weeks 3, 4, 8, 12, 16, 20 and 24
  The following laboratory variables will be measured and evaluated:
  Albumin, total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma glutamyl transferase (GGT), alkaline phosphatase (AP).
Changes in the profile of 80 different immunomodulatory cytokines at Weeks 3, 4, 8, 12, 16, 20 and 24 | Weeks 3, 4, 8, 12, 16, 20 and 24
  Fluorescence based analysis of 80 different immunomodulatory cytokine parameters in the patient's serum samples as assessed by a 80plex Human Cytokine Antibody Array Kit.
Changes in dialytic treatment until Week 24 | Between Screening and Week 24
  For patients with dialysis prior to Screening: Time to first dialysis after first IMP administration and time to last dialysis after first IMP administration until Week 24 will be assessed.
  For patients with no dialytic treatment prior to Screening the overall diaylsis timespan from first dialysis after first IMP administration until last dialysis will be measured.
Time to respiratory failure after first IMP administration until Week 24 | Between Day 0 (after first IMP administration) and Week 24
  Timespan to respiratory failure after first IMP administration until Week 24 will be measured.
Duration of the initial hospital stay | Between Screening and Week 24
  Initial hospitalisation time will be evaluated.
Duration of initial intensive care stay | Between Screening and Week 24
  The duration of initial intensive care stay will be evaluated.
Optional: Evaluation of liver biopsy (necrosis quantification) | Between Week 8 and Week 24
  Extent of necrosis will be quantified by the pathologist of the clinical trial center.
Physical examination at Week 24 | Week 24
  A physical body examination (e.g. general appearance, thyroid, head, lungs and thorax, ears, cardiovascular system, eyes, abdomen, nose-mouth-throat, musculoskeletal system, skin, extremities, lymph nodes, neurological system) will be performed and abnormal physical examination results will be evaluated and reported as AEs.
Vital signs at Week 24: Body temperature | Week 24
  Body temperature will be measured.
Vital signs at Week 24: Blood pressure | Week 24
  Blood pressure will be measured.
Vital signs at Week 24: Heart rate | Week 24
  Heart rate will be measured.
Vital signs at Week 24: Respiratory rate | Week 24
  Respiratory rate will be measured.
Hematological laboratory parameters at Week 24 | Week 24
  The hematological laboratory values for "hemoglobin, hematocrit, red blood cell count, white blood cell count with differential, platelet count" will be measured.
Clinical chemistry parameters at Week 24 | Week 24
  The clinical chemistry values for "sodium, potassium, calcium, urea, creatinine, albumin, total bilirubin, alanine aminotransferase, aspartate aminotransferase, gamma glytamyl transferase, alkaline phosphatase, CRP" will be measured.
Coagulation parameter "factor V" at Week 24 | Week 24
  The coagulation value for "factor V" will be measured.
Coagulation parameter "INR" at Week 24 | Week 24
  The coagulation value for "INR" will be measured.
Overall survival at Week 24 and at Month 24 | Week 24, Month 24
  Overall survival at Week 24 and at Month 24 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Ebert, Prof. Dr., Principal Investigator — Med. Fakultät Mannheim der Universität Heidelberg, II. Med. Klinik, Germany
Locations (5):
- Germany (5):
  - Universitätsklinikum Carl-Gustav-Carus an der TU Dresden, Medizinische Klinik I, Dresden
  - Universitätsklinikum Essen, Klinik für Gastroenterologie und Hepatologie, Medizinisches Forschungszentrum, Essen
  - Universitätsklinikum Frankfurt, Medizinische Klinik 1, Sektion Translationale Hepatologie, Frankfurt
  - Universitätsklinikum Magdeburg A.ö.R., Medizinische Fakultät der Otto-von-Guericke-Universität, Magdeburg
  - Medizinische Fakultät Mannheim der Universität Heidelberg, II. Medizinische Klinik, Mannheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerstan A, Niebergall-Roth E, Esterlechner J, Schroder HM, Gasser M, Waaga-Gasser AM, Goebeler M, Rak K, Schrufer P, Endres S, Hagenbusch P, Kraft K, Dieter K, Ballikaya S, Stemler N, Sadeghi S, Tappenbeck N, Murphy GF, Orgill DP, Frank NY, Ganss C, Scharffetter-Kochanek K, Frank MH, Kluth MA. Ex vivo-expanded highly pure ABCB5+ mesenchymal stromal cells as Good Manufacturing Practice-compliant autologous advanced therapy medicinal product for clinical use: process validation and first in-human data. Cytotherapy. 2021 Feb;23(2):165-175. doi: 10.1016/j.jcyt.2020.08.012. Epub 2020 Oct 1. PMID 33011075